CLINICAL TRIAL: NCT01184274
Title: A Phase I Study of SB939 in Pediatric Patients With Refractory Solid Tumours and Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Collaborators: S*BIO (Industry)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I203
Record Dates: First submitted 2010-08-17; First posted 2010-08-18 (Estimated); Last update posted 2023-08-04 (Actual); Status verified 2020-04

CONDITIONS: Leukemia; Solid Tumours
MeSH Terms: conditions — Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SB939 (Experimental)
  Interventions: Drug: SB939

INTERVENTIONS:
Drug: SB939 — Dose Levels for Part A
  -1 - 20mg/m2 - oral - Every other day three times/week1 for three consecutive weeks, followed by one week off-dosing
  1. (starting dose) 25mg/m2 - oral - Every other day three times/week1 for three consecutive weeks, followed by one week off-dosing
  2. - 35mg/m2 - oral - Every other day three times/week1 for three consecutive weeks, followed by one week off-dosing
  3. - 45mg/m2 - oral - Every other day three times/week1 for three consecutive weeks, followed by one week off-dosing
  4+ - Previous level + 10mg/m2 - oral - Every other day three times/week1 for three consecutive weeks, followed by one week off-dosing

SUMMARY:
This research is being done because SB939 has been shown to shrink tumours in animals and in some people and seems promising, but we are not sure if it can offer better results than standard treatment.

DETAILED DESCRIPTION:
In Part A of this study, SB939 was given to children with solid tumours. The purpose of Part A of this study is to ind the highest dose of a new drug SB939 that can be giben to children without causing very severe side effects that are tolerable.

In Part B of this study, SB939 will be given to children with leukemia. The purpose of Part B, is to see whether the dose that was determined to be the best dose for patients with solid tumours is also the best dose for children with leukemia.

In Part C of this study, SB939 will be given together with 13-cis-retinoic acid. The purpose of Part C, is to see whether the SB939 dose that was determined to be the best dose in Part A is also the best dose when given in combination with 13-cis-retinoic acid.

ELIGIBILITY:
Inclusion Criteria:

* Patients in all parts of the study must have histological verification of malignancy at either original diagnosis or relapse.

  * For Part A, patients must have recurrent or refractory solid tumours, lymphoma or CNS tumours (excluding diffuse intrinsic pontine gliomas).
  * For Part B, patients must have recurrent or refractory leukemia.
  * For Part C, patients must have one of the following diagnoses: neuroblastoma, or medulloblastoma / CNS primitive neuroectodermal tumour (PNET).

Disease Status

* Patients with solid tumours must have either measurable or evaluable disease (defined by a positive nuclear scan such as bone scan or metaiodobenzylguanidine (MIBG) scan. For part C only, in the case of neuroblastoma, if a lesion is isolated and /or previously irradiated and stable, a proven positive biopsy will be required to be eligible.
* Patients with refractory or relapsed leukemia must have greater than 25% blasts in bone marrow (M3 bone marrow); active extramedullary disease may also be present. Patients with leptomeningeal disease are not eligible.

Therapeutic Options:

The patient's current disease state must be one for which there is no known curative therapy or therapy proven to prolong survival with an acceptable quality of life.

Prior Systemic Therapy

Patients must have recovered from the acute effects of prior chemotherapy, immunotherapy or radiotherapy prior to study entry as follows:

* At least 3 weeks from completion of myelosuppressive chemotherapy, biologic agents or other investigational cancer treatment
* At least 7 days from completion of therapy with a growth factor
* At least 6 weeks from hematopoietic stem cell rescue following myeloablative therapy
* Post allogeneic hematopoietic transplant patients are eligible, but must have no evidence of active graft vs. host disease
* At least 2 weeks from completion of local palliative XRT (small port)
* At least 3 months must have elapsed if prior total body irradiation, craniospinal XRT or if ≥ 50% radiation of pelvis
* At least 6 weeks must have elapsed if other substantial bone marrow irradiation
* At least 6 weeks from prior MIBG therapy Age > 12 months and ≤ 18 years at the time of study entry. Performance Status: Karnofsky ≥ 60% for patients > 10 years; Lansky ≥ 50 for patients ≤ 10 years.

For Patients with Solid Tumours (Parts A and C):

* Absolute neutrophil count (ANC) ≥ 1.0 x 10 (power of 9)/L
* Platelets ≥100 x 10(power of 9)/L
* Hemoglobin ≥ 80 g/L

For Patients with Leukemia (Part B only)

* No minimum absolute neutrophil count
* Platelet count ≥ 20 x 10 (power of 9)/L (may receive transfusion)
* Hemoglobin ≥ 80 g/L (may receive transfusion)
* serum creatinine ≤ 1. 5 x upper limit of normal for age or
* measured GFR ≥ 70 mL/min/1.73 m2
* LVEF by ECHO or MUGA Scan within normal institutional limits
* QTc ≤ 450 msec

  * AST and ALT ≤ 5.0 x upper limit normal for age
  * bilirubin ≤ 1.5 x upper limit normal for age

Additional Criteria For Part C Of The Study

* Skin toxicity (excluding alopecia) ≤ Grade 1
* Serum triglycerides (fasting) < 3.4 mmol/L
* Negative urine dipstick for protein OR < 1000 mg protein/24 hour urine collection
* No evidence of gross hematuria

Patient or guardian consent must be obtained on all patients according to local Institutional and/or University Human Experimentation Committee requirements.

Patients registered on this trial must be treated and followed at the participating centre.

Protocol treatment to begin within five working days of patient registration.

Exclusion Criteria:

* Cardiac Exclusions. Patients with a pathologic cardiac arrhythmia requiring active treatment. Patients with a history of arrhythmia must be > 12 months since last treatment with no recurrence of arrhythmia in the interval.
* Inability To Take Oral Medication. Patients must be able to take oral medication and have no gastrointestinal abnormalities (e.g. bowel obstruction or previous gastric resection) which would lead to inadequate absorption of SB939.
* Known HIV, hepatitis B or hepatitis C infections.
* Current treatment with agents with a known risk of Torsades de Pointes http://torsades.org (list #1).
* Pre-existing peripheral neuropathy ≥ grade 3.
* There is no available information regarding human fetal or teratogenic toxicities related to SB939. 13-cis-retinoic acid is known to be teratogenic. Pregnancy tests must be obtained in girls who are post menarchal. Males or females of reproductive potential may not participate unless they have agreed to an effective contraceptive method. Pregnant or breast feeding females will not be entered on this study due to the potential fetal and teratogenic adverse events.

Ages: 12 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2010-10-01 (Actual); Primary Completion 2012-04-12 (Actual); Study Completion 2014-01-16 (Actual)

PRIMARY OUTCOMES:
Part A: Maximum Tolerated Dose and RP2D in solid tumours | 24 months
  Part A: patients must have recurrent or refractory solid tumours, lymphoma or CNS tumours (excluding diffuse intrinsic pontine gliomas)
  Purpose is to determine recommended phase II dose (RP2D) of oral SB939 in pediatric patients with solid tumours, with SB939 administered at a starting dose of 25 mg/m2 (70% of the adult recommended phase II dose), and given orally every other day three times / week (e.g. Monday / Wednesday /Friday OR Tuesday / Thursday / Saturday) for three consecutive weeks, followed by one week off-dosing.
Part B: Tolerability | 24 months
  Part B: patients must have recurrent or refractory leukemia
  Tolerability of the solid tumour RP2D in patients with recurrent or refractory leukemia once the RP2D has been established in solid tumours.
Part C: Recommended Phase 2 Dose (RP2D) and Tolerability | 24 months
  Part C: patients must have neuroblastoma, or medulloblastoma/CNS primitive neuroectodermal tumour (PNET)
  RP2D of oral SB939 in combination with a fixed dose of 13-cisretinoic acid in children with refractory or recurrent neuroblastoma, medulloblastoma / CNS neuroectodermal tumour (PNET), using the recommended dose determined in Part A of this study.
Pharmacokinetics | 24 months
  characterize the pharmacokinetics of SB939 in a pediatric population

SECONDARY OUTCOMES:
Anti-tumour activity | 24 months
  antitumour activity of SB939 in pediatric tumours when given as a single agent, and when given in combination with 13-cis-retinoic acid.

CONTACTS AND LOCATIONS:
Overall Officials: Sylvain Baruchel, Study Chair — Hospital for Sick Children, Toronto Ontario Canada
Locations (8):
- Canada (8):
  - Alberta Children's Hospital, Calgary, Alberta
  - Stollery Children's Hospital, Edmonton, Alberta
  - Children's and Women's Health Centre of BC Branch, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Izaak Walton Killam (IWK) Health Centre, Halifax, Nova Scotia
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - CHU Sainte-Justine, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zorzi AP, Bernstein M, Samson Y, Wall DA, Desai S, Nicksy D, Wainman N, Eisenhauer E, Baruchel S. A phase I study of histone deacetylase inhibitor, pracinostat (SB939), in pediatric patients with refractory solid tumors: IND203 a trial of the NCIC IND program/C17 pediatric phase I consortium. Pediatr Blood Cancer. 2013 Nov;60(11):1868-74. doi: 10.1002/pbc.24694. Epub 2013 Jul 25. PMID 23893953